CLINICAL TRIAL: NCT05679258
Title: A Phase I Study to Compare the Pharmacokinetic Characteristics, Safety, Tolerability, and Immunogenicity (Randomized, Double-blind, Parallel Controlled) of HLX15 With Daratumumab Injection in Healthy Chinese Male Subjects
Brief Title: A Study to Compare the PK , Safety, Tolerability, and Immunogenicity of HLX15 With Daratumumab in Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX15-001
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
Keywords: pharmacokinetics; CD38; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX15 group (Experimental): Recombinant anti-CD38 fully human monoclonal antibody injection developed by Shanghai Henlius Biotech, Inc.
  Interventions: Drug: HLX15
- US-sourced DARZALEX® group (Active Comparator): Daratumumab injection
  Interventions: Drug: US-sourced DARZALEX®
- CN-sourced DARZALEX® group (Active Comparator): Daratumumab injection
  Interventions: Drug: CN-sourced DARZALEX®
- EU-sourced DARZALEX® group (Active Comparator): Daratumumab injection
  Interventions: Drug: EU-sourced DARZALEX®

INTERVENTIONS:
Drug: HLX15 — A single dose (8 mg/kg) of HLX15 via intravenous infusion.
  Other Names: Recombinant anti-CD38 fully humanized monoclonal antibody injection
  Arms: HLX15 group
Drug: US-sourced DARZALEX® — A single dose (8 mg/kg) of US-sourced DARZALEX® via intravenous infusion.
  Other Names: Daratumumab Injection
  Arms: US-sourced DARZALEX® group
Drug: CN-sourced DARZALEX® — A single dose (8 mg/kg) of CN-sourced DARZALEX® via intravenous infusion.
  Other Names: Daratumumab Injection
  Arms: CN-sourced DARZALEX® group
Drug: EU-sourced DARZALEX® — A single dose (8 mg/kg) of EU-sourced DARZALEX® via intravenous infusion.
  Other Names: Daratumumab Injection
  Arms: EU-sourced DARZALEX® group

SUMMARY:
Phase I Study to Compare the Pharmacokinetic Characteristics, Safety, Tolerability, and Immunogenicity (Randomized, Double-blind, Parallel Controlled) of HLX15 with Daratumumab Injection in Healthy Chinese Male Subjects

DETAILED DESCRIPTION:
This study contains two parts. Part I of the study is a single-center, randomized, open-label, 2-arm, parallel-controlled phase Ia study to compare the PK characteristics, safety, tolerability, and immunogenicity of HLX15 and daratumumab infusion (DARZALEX®, CN-sourced) in healthy Chinese male subjects.

A total of 24 healthy Chinese male subjects will be enrolled in this part and randomized to the HLX15 group or the CN-sourced DARZALEX® group in a 1:1 ratio, with 12 subjects in each group. The subjects will receive a single dose (8 mg/kg) of HLX15 or CN-sourced DARZALEX® via intravenous infusion.

There is a safety run-in period in the early stage of the study to investigate the safety and tolerability of HLX15 in healthy Chinese male subjects. Another 3-6 subjects will be enrolled to receive the investigational product HLX15 and safety observation will be conducted for 1 week. The Safety Review Committee (SRC) will decide whether to adjust the subsequent study plan based on the safety and tolerability data after administration.

Part II of the study is a multicenter, randomized, double-blind, 3-arm, parallel-controlled phase Ib study to compare similarity of the PK characteristics, safety, tolerability, and immunogenicity of HLX15 and daratumumab infusion (DARZALEX®, US-sourced; DARZALEX®, CN-sourced) in healthy Chinese male subjects.A total of 204 healthy Chinese male subjects are planned to be enrolled in this part and randomly assigned in a 1:1:1 ratio to the HLX15 group, the US-sourced DARZALEX® group, or the CN-sourced DARZALEX® group, with 68 subjects in each group. The subjects will receive a single dose (8 mg/kg) of HLX15, US-sourced DARZALEX®, or CN-sourced DARZALEX® via intravenous infusion.This part may be adjusted according to the results of Part I, including sample size and sampling time points

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 60 years at the time of signing the informed consent form (ICF);
2. Sex: male;
3. Body weight and body mass index (BMI): 18.5 kg/m2 ≤ BMI < 28 kg/m2; body weight ≥ 55 kg;
4. The subject should be judged by the physician to be in good general health according to the results of medical history, physical examination, vital signs, ECG examination, laboratory tests, etc. (normal or abnormal without clinical significance);
5. The subject should be a voluntary participant who has understood and signed the ICF.

Exclusion Criteria:

1. Subjects who may have diseases that affect their safety or affect the study results, including but not limited to cardiovascular, respiratory, endocrine, metabolic, renal, hepatic, gastrointestinal tract, skin, infection, malignant tumor, hematologic, skeletal, genitourinary, nervous system/ psychiatric or functional disorders, which are judged as clinically significant by the investigator;
2. With acute, chronic, or latent infectious diseases within 1 month before administration;
3. With known immune system diseases (autoimmune diseases and immunodeficiency diseases), including but not limited to autoimmune hemolytic anemia;
4. Has experienced a recent single dermatomal herpes zoster eruption within 6 months before administration;
5. Has a history of multi-dermatomal herpes zoster or central nervous system (CNS) herpes zoster during the screening period or before;
6. Positive for indirect antiglobulin test (Indirect Coombs test);
7. Use of monoclonal antibody, cell therapy, etc. within 6 months before administration, or daratumumab or its analogues or drugs targeting CD38 before administration;
8. Use of any medication, including prescription drugs, over-the-counter (OTC) drugs, and Chinese herbal medicines, within 2 weeks before administration;
9. History of drug or food allergy, including allergy to any drug or drug excipient used in the study;
10. Fear of needles or blood, or difficulty in venous blood collection (history of difficult blood collection or corresponding symptoms and signs, unable to tolerate venipuncture);
11. History of blood donation or total blood loss of 200 mL or more within 3 months before administration;
12. Participants in clinical trials of any other drug or device within 3 months (or 5 half-lives of the corresponding investigational product if the half-life of the drug is long (5 half-lives > 3 months)) before administration;
13. Major surgery within 3 months before signing the ICF;
14. Positive for hepatitis B virus (HBsAg or HBcAb-positive) antibodies, hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV), or treponema pallidum antibodies (Anti-TP);
15. History of drug abuse or substance abuse, or positive in urine drug screening;
16. Patients who have been vaccinated with attenuated or live virus vaccine (such as Bacille Calmette-Guérin, BCG) or viral vector vaccine within 12 months before the first dose, or who plan to be vaccinated with such vaccines within 12 months after administration;
17. Patients who have been vaccinated with vaccines other than the above attenuated or live viral vaccines and viral vector vaccines within 1 month before the first dose, such as inactivated vaccines and recombinant subunit vaccines;
18. Male subjects with partners of childbearing potential who have a plan to father a child and/or donate sperm from signing of ICF through 3 months after administration, do not agree to abstain completely from sexual intercourse, or plan to use a contraceptive method that is not acceptable to the investigator (unacceptable methods of contraception include: i. periodic abstinence <such as calendar method, ovulation method, basal body temperature method, post-ovulation safety period method, etc.>, withdrawal, etc.; ii. medical contraceptive measures such as oral contraceptives, contraceptive injections, contraceptive patches, subcutaneous implantation, intrauterine hormone contraceptive devices, local contraceptives such as spermicides, etc.);
19. Subjects with any other conditions that, in the judgment of the investigator, are ineligible for participation in the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to infinity (AUC0-inf). | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

SECONDARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to the last measurable concentration (AUC0-t); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Maximum (peak) serum drug concentration (Cmax); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to reach maximum (peak) serum drug concentration (Tmax); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Volume of distribution during the terminal phase (Vz); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Elimination half-life (t1/2); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Total clearance (CL); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Percentage of area under serum concentration-time curve obtained by extrapolation (%AUCex). | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

OTHER OUTCOMES:
Adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal vital signs | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal physical examination findings; | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal Laboratory tests results (hematology, serum chemistry, and urinalysis); | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal 12-lead ECG readings. | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Incidence rate of anti-drug antibody (ADA) and NAb | Up to Day 91
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Sir Run Run Hospital, Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No